CLINICAL TRIAL: NCT01122823
Title: Evaluation of the Online Chronic Disease Self-Management Project at Group Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2008-Innov-4
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Chronic Conditions
Keywords: Chronic Disease Self-Management Program (CDSMP)
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- On-line workshop (Experimental): The online CDSMP is an internet-based program for people with 1 or more chronic conditions. It's built on self-efficacy theory, facilitated by lay leaders, and uses a curriculum emphasizing problem solving, decision making, and confidence building in weekly sessions over six weeks. It addresses generic topics and skills relevant to managing any chronic condition, including: action plans; problem solving; nutrition; exercise; fatigue; breathing; managing medications; managing stress and emotions; working with health care providers. The structure includes: 1) password-protected, interactive web-based instruction; 2) web-based bulletin board discussion groups to enable participatory learning and support; 3) and a reference book that contains the program content and supplemental information.
  Interventions: Behavioral: chronic disease self-management program (online)

INTERVENTIONS:
Behavioral: chronic disease self-management program (online) — The online CDSMP is an internet-based program for people with 1 or more chronic conditions. It's built on self-efficacy theory, facilitated by lay leaders, and uses a curriculum emphasizing problem solving, decision making, and confidence building in weekly sessions over six weeks. It addresses generic topics and skills relevant to managing any chronic condition, including: action plans; problem solving; nutrition; exercise; fatigue; breathing; managing medications; managing stress and emotions; working with health care providers. The structure includes: 1) password-protected, interactive web-based instruction; 2) web-based bulletin board discussion groups to enable participatory learning and support; 3) and a reference book that contains the program content and supplemental information.
  Other Names: Healthier Living with Ongoing Health Problems; Chronic Disease Self-Management Program

SUMMARY:
The purpose of this study is to learn if Group Health members who participate in the online chronic disease self-management program will experience improved health outcomes, improved health care utilization, and lower costs.

DETAILED DESCRIPTION:
We will pilot an evidence-based online program for chronic disease self-management that is modeled after the widely-replicated in-person Chronic Disease Self-management Program (CDSMP) developed at Stanford University.

The online CDSMP is an internet-based intervention for people with one or more chronic conditions. It is built on self-efficacy theory and is structured around a formal curriculum that emphasizes problem solving, decision making, and confidence building in weekly sessions over six weeks. The curriculum addresses generic topics and skills that are relevant to managing any chronic condition.

The program is structured around three components: 1) password-protected, interactive web-based instruction; 2) web-based bulletin board discussion groups to enable participatory learning and interaction; 3) and a reference book, Living a Healthy Life with Chronic Conditions, that contains the program content and supplemental information. It is facilitated by two trained lay moderators, at least one of whom has a chronic condition.

Piloting the online CDSMP allows Group Health to learn about and maximize the program's impact in the Group Health system before launching a full-scale program. Since web-based interventions are increasingly recognized as holding promise in health care, our learnings and recommendations will likely be applicable beyond this innovation. The pilot provides GH the opportunity to explore the following about the online CDSMP and web-based tools, in general:

1. Impact of the online CDSMP on participants' psychosocial and health status, health behaviors, and health service utilization
2. Efficient processes for incorporating the online CDSMP into existing operations through use of PDCA cycles
3. An understanding of demographic characteristics of members who are more likely to participate in an online self-management program than an in-person program
4. Effective recruitment and retention strategies
5. Feasibility of sustaining the program without external funding
6. Recommendations for successful implementation of future innovations that utilize web-based media, social networking technology, etc.

ELIGIBILITY:
Inclusion Criteria:

* Group Health member
* Have access to Group Health enhanced online services
* one or more chronic conditions or a caregiver of someone who fits that criteria
* 18 years of age or older

Exclusion Criteria:

* Not a Group Health member
* No access to Group Health enhanced online services
* No chronic conditions and not a caregiver of someone with a chronic condition
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
health outcomes | 6 months and 1 year after the intervention
  health status; self-efficacy; activities of daily living; symptomatology; mood; weight

SECONDARY OUTCOMES:
health care utilization | 6 months and 1 year after intervention
  number of physician visits, number of hospitalizations, number of nights in the hospital (all in past 6 months)
health behaviors | 6 months and 1 year after interventio
  physical activity; stress management; medication adherence; communication with health care team;

CONTACTS AND LOCATIONS:
Overall Officials: Judith Schaefer, MPH, Principal Investigator — Group Health Research Institute
Locations (1):
- Group Health Cooperative, Seattle, Washington, United States